CLINICAL TRIAL: NCT03334786
Title: An Open Label Study to Evaluate the Safety and Efficacy of FLX-787-ODT for Treatment of Fasciculations in the Tongue and One Appendicular Muscle in Adult Subjects With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Study to Evaluate Safety & Efficacy of FLX-787-ODT to Treat Fasciculations in Tongue and Appendicular Muscle in Adult Subjects With ALS
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Development of Current Formulation has Ceased
Sponsor: Flex Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLX-787-107
Record Dates: First submitted 2017-10-26; First posted 2017-11-07 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-04

CONDITIONS: Amyotrophic Lateral Sclerosis; Fasciculation
Keywords: ALS; Amyotrophic Lateral Sclerosis; Fasciculation; FLX-787
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Fasciculation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FLX-787-ODT (orally disintegrating tablet) (Experimental): Single dose
  Interventions: Drug: FLX-787-ODT

INTERVENTIONS:
Drug: FLX-787-ODT — Oral Disintegrating Tablet

SUMMARY:
The FLX-787-107 study will determine how well FLX-787-ODT works to reduce fasciculations in patients with Amyotrophic Lateral Sclerosis (ALS). The study will measure how often fasciculations occur, if tongue and muscle strength, speech, and swallowing are affected, and monitor any side effects that might develop while taking the investigational product. Participants will be assessed before and after taking a single dose of FLX-787-ODT. Approximately 15 people will take part in this study at one center in the United States. Participants will be in the study for a single clinic visit and receive a telephone call 7 days later to monitor for side effects.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of ALS diagnosis of less than 5 years.
* Greater than 6 fasciculations per minute noted at least in the tongue by clinical, ultrasound, or EMG evaluation.
* Normal oral cavity exam at screening.

Exclusion Criteria:

* Presence of clinically significant or unstable condition that would result in an increased risk of study participation or difficulty in interpretation of the study results.
* Tremor or other movement disorder that would interfere with recording.
* Presence of major gastrointestinal disorders, such as inflammatory bowel disease, diverticulitis, active peptic ulcer disease, or significant gastroesophageal reflux disease (i.e., not well-controlled on antacids or proton pump inhibitors), or oral or esophageal lesions/ulcers.
* Presence of laryngospasm or significant swallowing problems.
* Inability to tolerate a spicy sensation in the mouth or stomach.
* Actively using illicit drugs or history of chronic substance abuse within the past year prior to screening, including abuse of alcohol.
* Participated in a clinical study (except natural history studies without administration of an investigational product) within 30 days prior to screening.
* Pregnant, breastfeeding, or planning to become pregnant.
* Blood pressure of ≥160 mmHg systolic and/or ≥100 mmHg diastolic.
* Clinically significant abnormalities in laboratory findings (including screening complete electrolyte panel, complete blood count, liver function tests).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2018-08-23 (Actual); Study Completion 2018-08-23 (Actual)

PRIMARY OUTCOMES:
Change from Baseline of Diastolic Blood Pressure in mmHg | Prior to and within 3 hours following administration of investigational product on the single clinic visit
  Diastolic blood pressure collected before and after treatment
Change from Baseline of Systolic Blood Pressure in mmHg | Prior to and within 3 hours following administration of investigational product on the single clinic visit
  Systolic blood pressure collected before and after treatment
Change from Baseline in Heart Rate in beats per minute | Prior to and within 3 hours following administration of investigational product on the single clinic visit
  Heart rate collected before and after treatment
Change from Baseline in Respiration Rate in breaths per minute | Prior to and within 3 hours following administration of investigational product on the single clinic visit
  Respiration rate collected before and after treatment
Change from Baseline in Body Temperature in degrees Celsius or Fahrenheit | Prior to and within 3 hours following administration of investigational product on the single clinic visit
  Body temperature collected before and after treatment
Change from Baseline of Oral Cavity Examination | Prior to and twice within 4 hours following administration of investigational product on the clinic visit
  Oral Cavity Examination performed before and after treatment
Incidence of Treatment-Emergent Adverse Events | Prior to and following administration of investigational product on the clinic visit with AEs followed for 7 days after by telephone contact
  Adverse Event Information collected throughout the study

SECONDARY OUTCOMES:
Change from Baseline of Fasciculation Frequency | Prior to and twice within 4 hours following administration of investigational product on the clinic visit
  Fasciculations over time measured by ultrasound before and after treatment
Change from Baseline of Fasciculation Frequency | Prior to and twice within 4 hours following administration of investigational product on the clinic visit
  Fasciculations over time measured by EMG before and after treatment
Change from Baseline in Peak Tongue Strength in kPa by Iowa Oral Performance Instrument | Prior to and once within 4 hours following administration of investigational product on the clinic visit
  Peak Tongue Strength Measurements before and after treatment
Change from Baseline in Speech Assessments | Prior to and once within 4 hours following administration of investigational product on the clinic visit
  Timed Speech Assessments before and after treatment
Change from Baseline in Swallowing Assessments | Prior to and once within 4 hours following administration of investigational product on the clinic visit
  Timed Swallowing Assessments before and after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided